CLINICAL TRIAL: NCT06240611
Title: Isokinetic Assessment of Wrist Muscle Performance Among Egyptian Physical Therapy Students With Chronic Non-Specific Neck Pain
Brief Title: Isokinetic Assessment of Wrist Muscle Performance Among Medical Students With Neck Pain
Status: Completed | Type: Observational
Sponsor: Mohamed Mahmoud Refaey (Other)
Responsible Party: Sponsor-Investigator, Mohamed Mahmoud Refaey, Department of Biomechanics, Faculty of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: neck pain on wrist muscles
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
Keywords: Muscle Strength; Muscle Fatigue; Dynamometer; Wrist
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Control): A healthy matched volunteers' group (n = 23) between 18 and 23 years of age was included in this study. For students of both genders, the body mass index was not less than 18.5 and not more than 29.5, and there was no recent or previous musculoskeletal injury or pain.
- Group B (Experimental): Participants with CNSNP (n = 22) were between 18 and 23 years of age. Patients with CNSNP For students of both genders, the duration of the non-specific neck pain was more than 3 months (for the symptomatic group with no neurological manifestations and with referral from orthopedic surgeons by diagnosis of non-specific neck pain), and for matched students, they did not have any history of neck pain. The student's age ranges from 18 to 23 years. Neck pain intensity on the numerical Pain Rating Scale was between 3 and 8, and neck pain-related disability on the Neck Disability Index was between 5 and 14 points (10-28%) for mild disability and 15-24 points (30-48%) for moderate disability. The body mass index for students was not less than 18.5 and not more than 29.5.

SUMMARY:
PURPOSES:

1. To assess the effect of chronic non-specific neck pain on peak torque of wrist extensor and flexor muscles /body weight among Egyptian physical therapy students.
2. To assess the effect of chronic non-specific neck pain on extensor / flexor wrist ratio among Egyptian physical therapy students.
3. To assess the effect of chronic non-specific neck pain on wrist extensor and flexor muscles endurance among Egyptian physical therapy students.

DETAILED DESCRIPTION:
BACKGROUND:

Although it is widely acknowledged that chronic non-specific neck pain is linked to hand disability as previously studied on dentists and ministry of health care stuff, there is still a gap in illustrating the effect of chronic non-specific neck pain on Egyptian physical therapy students' functional ability of wrist in the upper limb. However, the assessment of extensor / flexor wrist strength ratio has only recently gained attention. Furthermore, there is limited research investigating the strength control ratio that incorporates both concentric and eccentric muscle actions, and additional scientific evidence is needed to establish the relationship between chronic non-specific neck pain and upper limb disability. This study will be conducted to set new assessment and rehabilitation goals. This will subsequently be translated into home therapy program, contributing to decrease the burden of neck pain economically and on health care management.

Our study aims to evaluate peak torque of wrist extensor and flexor muscle/ body weight and extensor / flexor wrist ratio and wrist extensor and flexor muscle endurance among Egyptian physical therapy students with non-specific neck pain. Torque results are adjusted for body weight and compared to normative data for the gender and activity specialty to determine whether the unaffected limb is strong enough to act as a reference for the afflicted limb also compared between right- and left-handed subjects.

HYPOTHESES:

* There will be no significant effect of chronic non-specific neck pain on peak torque of wrist extensor and flexor muscles /body weight.
* There will be no significant effect of chronic non-specific neck pain on extensor / flexor wrist ratio.
* There will be no significant effect of chronic non-specific neck pain on wrist extensor and flexor muscles endurance.

RESEARCH QUESTIONS:

* Does chronic non-specific neck pain affect wrist extensor and flexor muscles performance among Egyptian physical therapy students?
* Does chronic non-specific neck pain affect peak torque of wrist extensor and flexor muscles/ body weight among Egyptian physical therapy students?
* Does chronic non-specific neck pain affect extensor / flexor wrist ratio among Egyptian physical therapy students?
* Does chronic non-specific neck pain affect wrist extensor and flexor muscles endurance among Egyptian physical therapy students?

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Duration of neck pain (> 3 months)
* Age from 18 to 23 years
* The neck pain intensity is between 3 and 8 on the Numerical Pain Rating Scale
* Neck pain-related disability was between 5 and 14 points on the Neck Disability Index
* Body mass index from 18.5 to 29.5

Exclusion Criteria:

* Neurological conditions (i.e., Parkinson's disease, multiple sclerosis, head injury, peripheral neuropathy, stroke, or nerve root entrapment)
* Headache
* Cancer, infection, or any other illness symptoms.
* Trauma
* Cardiovascular problems or cerebrovascular insufficiency symptoms.
* Musculoskeletal disorder (i.e., joint replacement, amputation, physically limiting arthritis, contractures of fixed deformity, or muscular dystrophy)
* Orthopedic or neurological conditions such as fractures, surgeries on the upper limb or hand, carpal tunnel syndrome, De Quervain's syndrome, or diabetic mellitus
* Cervical spine spondylosis, disc prolapse, spinal stenosis, cervical fracture, etc.
* Any recent treatment for neck pain.
* Visual, auditory and speech problems
* Forward head posture.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were recruited from the physical therapy outpatients' clinics of Cairo University, and they were assigned into two groups (group A (control group) and group B (experimental group), with a sample size of approximately 44 participants and an anticipated 15% dropout rate (twenty-two in each group) calculated using the G Power test method.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the findings of isokinetic dynamometer between control and study groups | Baseline
  peak torque/body weight percentage between control and study groups
The difference between control and study groups in the findings of isokinetic dynamometer | Through study completion, an average of 5 months
  work fatigue index percentage between control and study groups
The correlation between neck pain and the findings of isokinetic dynamometer | Up to 5 months
  agonist/antagonist ratio percentage between control and study groups

CONTACTS AND LOCATIONS:
Overall Officials: Enas F Youssef, Dr, Study Chair — Department of Musculoskeletal Disorders Faculty of Physical Therapy Cairo University; Anees S Gheit, Dr, Study Director — Department of Biomechanics, Faculty of Physical Therapy Kafr El Sheikh University; Aya A Khalil, Principal Investigator — Department of Biomechanics, Faculty of Physical Therapy Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alreni AS, Harrop D, Gumber A, McLean S. Measures of upper limb function for people with neck pain: a systematic review of measurement and practical properties (protocol). Syst Rev. 2015 Apr 7;4:43. doi: 10.1186/s13643-015-0034-2. PMID 25875810
- [Result] Andrew D, Yielder P, Haavik H, Murphy B. The effects of subclinical neck pain on sensorimotor integration following a complex motor pursuit task. Exp Brain Res. 2018 Jan;236(1):1-11. doi: 10.1007/s00221-017-5103-4. Epub 2017 Oct 12. PMID 29026942
- [Result] Alsalameh AM, Harisi MJ, Alduayji MA, Almutham AA, Mahmood FM. Evaluating the relationship between smartphone addiction/overuse and musculoskeletal pain among medical students at Qassim University. J Family Med Prim Care. 2019 Sep 30;8(9):2953-2959. doi: 10.4103/jfmpc.jfmpc_665_19. eCollection 2019 Sep. PMID 31681674
- [Result] Ajimsha MS, Shenoy PD, Gampawar N. Role of fascial connectivity in musculoskeletal dysfunctions: A narrative review. J Bodyw Mov Ther. 2020 Oct;24(4):423-431. doi: 10.1016/j.jbmt.2020.07.020. Epub 2020 Jul 30. PMID 33218543
- [Result] de la Motte SJ, Gribbin TC, Lisman P, Murphy K, Deuster PA. Systematic Review of the Association Between Physical Fitness and Musculoskeletal Injury Risk: Part 2-Muscular Endurance and Muscular Strength. J Strength Cond Res. 2017 Nov;31(11):3218-3234. doi: 10.1519/JSC.0000000000002174. PMID 28796127
- [Result] Gane EM, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. The relationship between physical impairments, quality of life and disability of the neck and upper limb in patients following neck dissection. J Cancer Surviv. 2018 Oct;12(5):619-631. doi: 10.1007/s11764-018-0697-5. Epub 2018 May 16. PMID 29770954
- [Result] Ortego G, Lluch E, Herrero P, Boudreau SA, Domenech-Garcia V. Profiling and Association over Time between Disability and Pain Features in Patients with Chronic Nonspecific Neck Pain: A Longitudinal Study. J Clin Med. 2022 Feb 28;11(5):1346. doi: 10.3390/jcm11051346. PMID 35268437
- [Result] Stenner HT, Eigendorf J, Kerling A, Kueck M, Hanke AA, Boyen J, Nelius AK, Melk A, Boethig D, Bara C, Hilfiker A, Berliner D, Bauersachs J, Hilfiker-Kleiner D, Eberhard J, Stiesch M, Schippert C, Haverich A, Tegtbur U, Haufe S. Effects of six month personalized endurance training on work ability in middle-aged sedentary women: a secondary analysis of a randomized controlled trial. J Occup Med Toxicol. 2020 May 6;15:8. doi: 10.1186/s12995-020-00261-4. eCollection 2020. PMID 32391068

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT06240611/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Results of Agonist to Antagonist Ratio in Both Group (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT06240611/SAP_001.pdf
  • Statistical Analysis Plan: Results of Peak torque to Body weight in Both Group (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT06240611/SAP_002.pdf
  • Statistical Analysis Plan: Results of Work Fatigue in Both Group (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT06240611/SAP_003.pdf